## **Study title**

A DOUBLE-BLIND, RANDOMISED, PLACEBO-CONTROLLED PHASE I TRIAL TO INVESTIGATE SAFETY, TOLERABILITYAND PHARMACOKINETICS OF SINGLE ASCENDING TOPICAL DOSES OF GZ21T IN HEALTHY VOLUNTEERS

**NCT Number** 

NCT06888362

**Statistical Analysis Plan** 

v4.0; 28APR2025

Final v4.0; 28APR2025

Statistical Analysis Plan

SAP version and date

EU Trial No. 2024-512893-86-00

Investigational medicinal product GZ21T

Trial code A24-0001

Protocol version and date Final v2.0; 20NOV2024

A DOUBLE-BLIND, RANDOMISED, PLACEBO-CONTROLLED PHASE I TRIAL TO INVESTIGATE SAFETY, TOLERABILITYAND PHARMACOKINETICS OF SINGLE ASCENDING TOPICAL DOSES OF

**GZ21T IN HEALTHY VOLUNTEERS** 

Sponsor Ankh Life Sciences

Sponsor signatory

CTC biostatistician

Clinical Trial Consultants AB (CTC) Dag Hammarskjölds väg 10B SE-752 37 Uppsala, Sweden

This Statistical Analysis Plan is the property of Ankh Life Sciences and is a confidential document. It is not to be copied or distributed to other parties without written approval from Ankh Life Sciences.


 Table 1
 SAP version history

| SAP<br>version | Approval date | Description of changes |
|---|---|---|
| 1.0,<br>original<br>version | 04OCT2024 | |
| 2.0 | 28JAN2025 | The SAP was updated in accordance with the changes in the clinical trial protocol (CTP) v2.0 to include an additional part (Part B). This part consists of 1 cohort (3 participants), with the option to include up to 2 additional cohorts of 3 participants each, in order to evaluate the optimum amount of cream to be applied to a given body area (dose/area). |
| 3.0 | 05JAN2025 | Updated Sections 9.1.7 and 10.2.2.7 regarding the presentation of "time until adequate abruption" based on how the data is collected in the eCRF. |
| 4.0 | 28APR2025 | <ul> <li>Updated</li> <li>Section 7 to include full CDSIC compliance.</li> <li>Section 9.3.3 and Tables CM1 to CM4 to use WHODrug coding instead of ATC coding</li> <li>Changed CTC biostatistician</li> </ul> |


#### 1 SIGNATURES





Sponsor signatory



## 2 TABLE OF CONTENTS

| 1 | SIG | NATURES | 3 |
|---|-------|----------------------------------------------------|------|
| 2 | TAl | BLE OF CONTENTS | 4 |
| 3 | LIS | T OF ABBREVIATIONS AND DEFINITION OF TERMS | 6 |
| 4 | INT | RODUCTION | 8 |
| | 4.1 | Trial design | 8 |
| | 4.2 | Trial objectives and endpoints | 9 |
| | 4.3 | Randomisation (Part A) | . 11 |
| | 4.4 | Participant replacement | . 11 |
| | 4.5 | Blinding | . 11 |
| 5 | STA | ATISTICAL AND ANALYTICAL PLANS | . 12 |
| | 5.1 | Sample size calculation and number of participants | . 12 |
| | 5.2 | Definition of analysis sets | . 12 |
| | 5.3 | Compliance | . 12 |
| | 5.4 | Definition of baseline | . 12 |
| | 5.5 | Rounding principles | . 12 |
| | 5.6 | Handling of dropouts, missing data and outliers | . 13 |
| 6 | CH | ANGES FROM THE CLINICAL TRIAL PROTOCOL | . 14 |
| 7 | CLI | INICAL DATABASE PROCESSING | . 15 |
| | 7.1 | General information | . 15 |
| | 7.1. | 1 CDISC Compliance | . 15 |
| | 7.2 | Database modeling of trial design | . 16 |
| 8 | STA | ATISTICAL DELIVERABLES | . 18 |
| 9 | STA | ATISTICAL METHODOLOGY | . 19 |
| | 9.1 | Analysis of the primary endpoints | . 19 |
| | 9.1. | 1 Adverse events | . 19 |
| | 9.1.2 | 2 Local tolerability | . 19 |
| | 9.1. | 3 Vital signs | . 19 |
| | 9.1.4 | 4 Electrocardiogram | . 19 |
| | 9.1. | 5 Safety laboratory | . 19 |
| | 9.1.0 | 6 Physical examinations | . 20 |
| | 9.1. | 7 Cream absorption (Part B) | . 20 |
| | 9.2 | Analysis of secondary endpoints | . 20 |
| | 9.2. | Pharmacokinetic analysis (Part A) | . 20 |
| | 9.3 | Description of trial population | . 22 |
| | 9.3. | 1 Disposition | . 22 |

## **Ankh Life Sciences Limited**

| | Statistical Analysis Plan A24 | -0001 Final v4.0 |
|---|---|---|
| 9.3.2 | Demographics and baseline characteristics | 23 |
| 9.3.3 | Medical/surgical history and prior/concomitant medication | 23 |
| 9.3.4 | Investigational medicinal product use | 23 |
| 10 DA | ATA DISPLAY PLAN | 24 |
| 10.1 | Γable of contents DDP | 24 |
| List of table | es | |
| Гable 1 | SAP version history | 2 |
| Γable 2 | Trial objectives and endpoints (Part A) | 9 |
| Гable 3 | Trial objectives and endpoints (Part B) | 10 |
| Гable 4 | Analysis sets | 12 |
| Γable 5 | Changes in the planned statistical analyses | 14 |
| List of figur | res | |
| Figure 1 | Trial design and proposed doses | 8 |
| Figure 2 | Schematic representation of the SDTM trial design (Part A) | 16 |
| Figure 3 | Schematic representation of the SDTM trial design (Part B) | 17 |

## 3 LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation | Explanation |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse event |
| ATC | Anatomical therapeutic chemical |
| AUC | Area under the plasma concentration vs. time curve |
| $\mathrm{AUC}_{0\text{-inf}}$ | AUC from 0 to infinity |
| AUC <sub>0-last</sub> | AUC from 0 to time of last measurable plasma concentration |
| BLQ | Below lower limit of quantification |
| BMI | Body mass index |
| CDISC | Clinical Data Interchange Standards Consortium |
| $C_{last}$ | Last observed plasma concentration |
| $C_{\text{max}}$ | Maximum observed concentration |
| CTC | Clinical Trial Consultants AB |
| CTP | Clinical trial protocol |
| CV | Coefficient of variation |
| DDP | Data display plan |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| FAS | Full analysis set |
| FDA | United States Food and Drug Administration |
| FIH | First-in-human |
| Geo | Geometric |
| IG | Implementation guide |
| IMP | Investigational medicinal product |
| lin | Linear |
| LLOQ | Lower limit of quantification |
| LS | Least square |
| MAD | Multiple-ascending dose |
| Max | Maximum |
| MedDRA | Medical dictionary for regulatory activities |
| Min | Minimum |
| NA | Not applicable/not available |
| NC | Not calculated |

| Abbreviation | Explanation |
|------------------|-----------------------------------------|
| NCA | Non-compartmental analysis |
| PK | Pharmacokinetic(s) |
| PKAS | PK analysis set |
| PT | Preferred term |
| SAD | Single-ascending dose |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Statistical analysis system |
| SD | Standard deviation |
| SDTM | Trial data tabulation model |
| SOC | System organ class |
| $T_{last}$ | Time of occurrence of C <sub>last</sub> |
| $T_{\text{max}}$ | Time of occurrence of C <sub>max</sub> |
| $T_{1/2}$ | Terminal elimination half-life |
| ULOQ | Upper limit of quantification |
| ULQ | Above upper limit of quantification |
| WHO | World Health Organization |

#### 4 INTRODUCTION

This SAP gives a detailed description of the planned statistical analysis for trial A24-0001.

#### 4.1 Trial design

This trial is a Phase I-trial divided into 2 parts. Part A is, double-blind, placebo-controlled, and designed to evaluate the safety, tolerability, and PK after topical administration of single ascending doses of GZ21T in healthy male and female volunteers. Part B is open-label and designed to evaluate the optimum amount of cream applied to a given body area (dose/area) of single doses of GZ21T in healthy volunteers.

In Part A, participants will receive a single topical application of GZ21T or placebo in 2 sequential cohorts (cohorts 1 and 2) followed by 2 cohorts starting in parallel (cohorts 3 and 4) with planned doses as follows:



In Part B, participants in cohort 1 will receive a single topical application of GZ21T. Based on the extent of the cream's absorption, up to 2 additional cohorts can be explored (optional cohorts 2 and 3). The maximum administered dose will not exceed

The trial design and the proposed dose levels are shown in Figure 1. Please see the CTP for additional details.

Figure 1 Trial design and proposed doses



The dose levels for Part A cohorts 2, 3 and 4 are tentative. The internal safety review committee will review the safety, tolerability and PK data prior to initiating cohort 2, cohorts 3 and 4. The dose levels for Part B, optional cohorts 2 and 3, will be based on the result from preceding cohorts. BSA=body surface area.

# 4.2 Trial objectives and endpoints

Table 2 Trial objectives and endpoints (Part A)

| Objectives | Endpoints | Assessments | Analysis | Data display<br>plan (DDP) |
|---|---|---|---|---|
| Primary | | | | |
| To evaluate the safety and tolerability of GZ21T after single | Frequency, severity and intensity of adverse events (AEs). | AE reporting and questioning | Descriptive statistics,<br>Section 9.1.1 | Section 10.2.2.1 |
| topical dose applications. | Local tolerability reactions: Erythema, swelling, pruritus, burning, blistering and urticaria, discolouration and dryness (Investigator's assessment 0-3 none/mild/moderate/severe). | Local tolerability reactions | Descriptive statistics,<br>Section 9.1.2 | Section 10.2.2.2 |
| | Clinically significant changes in vital signs, electrocardiograms (ECGs), safety laboratory | Blood pressure and pulse | Descriptive statistics,<br>Section 9.1.3 | Section 10.2.2.3 |
| | measurements (haematology, clinical chemistry, coagulation) and physical examination findings. | 12-lead ECG | Descriptive statistics,<br>Section 9.1.4 | Section 10.2.2.4 |
| | | Blood sampling for haematology, clinical chemistry and coagulation | Descriptive statistics,<br>Section 9.1.5 | Section 10.2.2.5 |
| | | Physical examinations | Descriptive statistics,<br>Section 9.1.6 | Section 10.2.2.6 |
| Secondary | | | | |
| To investigate the potential systemic exposure and pharmacokinetic (PK) properties of GZ21T after single | Plasma concentrations of GZ21T after single dose applications. | PK sampling and analysis | Descriptive statistics,<br>Section 9.2.1 | Section 10.2.3.1 |
| topical dose applications. | PK parameters after a single dose application (to be calculated if data permits): area under the plasma concentration curve from time 0 to infinity (AUC $_{inf}$ ), AUC from time 0 to the last measurable concentration (AUC $_{last}$ ), maximum plasma concentration (C $_{max}$ ), time to C $_{max}$ (T $_{max}$ ), terminal elimination half-life (T $_{1/2}$ ). | _ | | |

Table 3 Trial objectives and endpoints (Part B)

| Objectives | Endpoints | Assessments | Analysis | DDP |
|---|---|---|---|---|
| Primary | | | | |
| To investigate the optimum amount of cream applied to a given area (dose/area) after single topical dose applications. | Cream absorption after single dose applications. | Evaluation of cream absorption | Section 9.1.7 | Section 10.2.2.7 |

#### 4.3 Randomisation (Part A)

On Day 1 (Visit 2), participants in each cohort (Part A) were randomised in a 6:2 ratio to receive either GZ21T or placebo. Sentinel dosing was applied for the first 2 participants in each cohort who received either GZ21T or placebo as randomised.

#### 4.4 Participant replacement

Participants who were prematurely withdrawn from the trial for any reason except the occurrence of AEs assessed as possibly or probably related to the trial treatment may have been replaced.

## 4.5 Blinding

Part A of the trial is double-blinded. The allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.

Part B of the trial is open-label and therefore no blinding will be performed.

#### 5 STATISTICAL AND ANALYTICAL PLANS

#### 5.1 Sample size calculation and number of participants

No formal sample size calculation has been performed for this trial. The proposed sample size is considered sufficient to provide adequate information to meet the trial objectives.

Part A: Approximately 64 participants were planned to be screened to achieve 32 randomised participants (8 in each cohort).

Part B: Approximately 18 potential participants were planned be screened to achieve up to 9 included participants, 3 subjects per cohort.

## 5.2 Definition of analysis sets

The analysis sets defined for the trial are outlined in Table 4.

Table 4 Analysis sets

| Analysis set | Definition | Comment | Use of analysis set |
|---|---|---|---|
| Full analysis set (FAS) | All enrolled participants who received Participants will only receive 1 dose of IMP. Therefore, the phrase (as stated in | Part A and Part B:<br>Safety endpoints and<br>description of trial<br>population. | |
| Pharmacokinetic<br>analysis set (PKAS) | All randomised participants in Part A who received IMP and provided an evaluable plasma concentration profile, and who have no AEs or protocol deviations judged to affect the PK analysis. Individual PK values may be excluded from the analysis. | the CTP) "at least 1 dose of" before "IMP" is removed from the definitions to minimise confusion. | Part A: PK endpoints. |

#### 5.3 Compliance

All IMP were administered at the trial site under medical supervision to ensure compliance.

#### **5.4** Definition of baseline

Baseline is defined as the last non-missing data collection point prior to the administration of IMP.

#### 5.5 Rounding principles

Generally, no rounding of data will be done prior to calculating statistics. However, if reported data contains more than 8 significant digits it will be rounded to 8 significant digits in the database.

In statistical output and descriptive summaries, the following principles will be used:

- Data will be presented as reported in input data in listings.
- Two (2) significant digits will be used for percentages (for example relative change from baseline).
- p-values and similar statistical output will be presented using 4 decimal places.
- Three (3) significant digits will be used for PK parameters when presenting min and max values in tables.

- Descriptive summaries (e.g., mean, SD, median etc.) of PK parameters will be presented with 4 significant digits.
- Descriptive summaries (e.g., mean, SD, median etc.) of all other numerical data will be presented with one extra decimal compared to reported input data.

#### 5.6 Handling of dropouts, missing data and outliers

Outliers will be included in summary tables and listings and will not be handled separately in any analyses. All collected data, even if not tabulated, will be listed. Generally, no imputation of data will be performed. However, when calculating statistics for PK plasma concentrations, concentrations under LLOQ will be replaced with LLOQ/2 if more than 50% of the values for a given time point are above LLOQ. Otherwise, no statistics will be calculated for that time point. For figures presenting individual PK concentrations, no imputation is performed for values under LLOQ. For imputation of PK plasma concentration below LLOQ with the purpose of calculating PK parameters, see Section 9.2.1.

Safety laboratory concentrations under LLOQ will be replaced with LLOQ/2 and concentrations over ULOQ will be replaced with ULOQ for the purpose of calculating descriptive statistics.

In case of missing start and stop times of AEs that cannot be investigated further, missing data will be imputed according to a worst-case scenario, i.e., start time will be imputed as the closest time point post first intake of IMP and end time as 23:59, resulting in the longest possible treatment emergent duration of the AE.

## 6 CHANGES FROM THE CLINICAL TRIAL PROTOCOL

Changes to the planned analyses and the timing of these are summarised in Table 5.

 Table 5
 Changes in the planned statistical analyses

| Change category | Timing of change | Description of change | Reason for change |
|---|---|---|---|
| Change in the SAP compared to the CTP | Prior to DBL | A minor change has been made to the phrasing of the definitions for FAS and PKAS. This change does not affect whether participants are included in the analysis sets or not. See Table 4 for details. | To minimise confusion. |
| | | In section 9.1.1, definitely related AEs has been added to the definition of causally related AEs, which is missing from sections 11.3.1.11 and 17.6.1 of the CTP. | "Definitely related" was<br>missing from the AE<br>definitions in sections<br>11.3.1.11 and 17.6.1 of the<br>CTP |
| | | Frequency tables for safety laboratory interpretations have been added. | To provide a better overview of the safety laboratory data. |
| | | The overall/total column has been removed from all safety tabulations, except for AEs and LTs. | Redundant information. |

#### 7 CLINICAL DATABASE PROCESSING

#### 7.1 General information

The clinical database is processed and generated according to The Clinical Data Interchange Standards Consortium (CDISC). CDISC is a Standard Developing Organization which develops and publishes standards to normalise the structure of clinical trial data and thereby simplify submissions to and reviews by authorities such as the Food and Drug Administration (FDA).

The CDISC standards for clinical studies are the Trial Data Tabulation Model (SDTM) and the Analysis Data Model (ADaM). The trial data will be structured into a database model reflecting the SDTM and will be compliant to SDTM Implementation Guide (SDTM-IG) version 3.3. The data used for statistical analysis will be structured to reflect the ADaM and be compliant to ADaM Implementation Guide (ADaM-IG) version 1.3.

Data values are collected according to, or mapped into, controlled terminology codelists defined by CDISC, whenever possible. The codelists are updated quarterly at CTC and the latest version available at trial start will be used. As per default, controlled terminology codelists will be used in all tables, listings, and figures. Custom codelists for test or parameter names will be used if applicable upon Sponsor's request, to align with protocol texts, or to adhere to other standard naming conventions (e.g., PK parameter name "Tmax" will be used instead of the CDISC term "Time of CMAX"). These custom codelists will be mapped in the "Parameter Name" field in the ADaM structure, while the CT will be kept in the SDTM predecessor fields to provide traceability back to CDISC codelists.

## 7.1.1 CDISC Compliance

The trial database will be CDISC compliant which means that the clinical database will be processed and generated according to CDISC standard. The database will be validated against SDTM and ADaM Validation rules using Pinnacle 21.

The following CDISC documentation will be generated:

- SDTM Data Definition Specification (also referred to as a Define -XML)
  - Define-XML transmits metadata that describes any tabular dataset structure and supports the interchange of dataset metadata for clinical research applications in a machine-readable format.
- ADaM Data Definition Specification (also referred to as a Define -XML)
  - Define-XML transmits metadata that describes any tabular dataset structure and supports the interchange of dataset metadata for clinical research applications in a machine-readable format.
- Annotated Electronic Case Report Form (eCRF)
  - Links the data collection fields used to capture trial data to the corresponding variables in the trial database. It enables the user to understand how the trial data were collected and to trace back from trial analysis results to the origin where it was collected.
- SDTM Reviewers' Guide
  - Intended to provide additional context and act as a single point of orientation for the SDTM datasets.
- ADaM Reviewers' Guide
  - Provides regulatory agency reviewers an orientation to the submitted analysis data in a consistent way and usable format.

### 7.2 Database modeling of trial design

The trial design is mapped to a SDTM trial design model containing the following structural components:

**EPOCH**: An interval of time in the planned conduct of a trial. An epoch is associated with a purpose (e.g., screening, randomisation, treatment, follow-up), and applies across all arms of the trial. Trial epochs follow a controlled terminology to represent the different trial parts (e.g., SCREENING, TREATMENT [X], FOLLOW-UP)

**ELEMENT**: Building blocks used to build up the entire trial length for all participants. Information on ELEMENTs is extracted from the trial design and schedule of events in the protocol. ELEMENTs are defined to span the entire trial without gaps. One EPOCH may contain one or several ELEMENTs. All ELEMENTs must have transition rules in accordance with the protocol to determine start and end.

**ARM**: Participants are allocated to trial arms depending on the trial design, either by randomisation or other allocation processes defined in the trial protocol. ARMs are defined as the total number of planned ways a participant can go through the trial (unique combination of trial ELEMENTs). All ARMs must contain a unique sequence of ELEMENTs.

**VISIT**: Trial visits are defined as planned timepoints during the trial where trial data is collected. A visit can be performed in clinic, by off-site contact with trial personnel (phone call, video conference or similar), or by participant initiated recordings of data. The visit schedule is extracted from protocol and eCRF design.

A schematic representation of the SDTM trial design is presented in Figure 2. Replace the figure below with a relevant version for the trial.





## 8 STATISTICAL DELIVERABLES

The following items will be delivered:

- Statistical analyses, summary tables, listings and figures as described under Section 10.
- Clinical trial database delivered as a SAS-export file and Excel files.

#### 9 STATISTICAL METHODOLOGY

All collected data will be listed by part, participant, cohort and treatment, and, where applicable, by assessment time.

The data for participants receiving placebo will be presented pooled across groups.

Details on statistical analyses and descriptive summaries are specified below.

All statistical analyses and descriptive summaries will be performed using SAS version 9.4 (SAS institute, Cary, NC).

PK parameters will be calculated by Non-Compartmental Analysis (NCA) using the software Phoenix WinNonlin® version 8.3 (Certara, U.S.A).

#### 9.1 Analysis of the primary endpoints

#### 9.1.1 Adverse events

An overview of all AEs, including SAEs, intensity, relationship to IMP, and deaths will be presented by part, cohort treatment, and overall. The incidence of AEs and SAEs will be summarised by SOC and PT by treatment, cohort and overall. A summary of any treatment-related (probably/possibly/definitely related) AEs will be summarised by SOC and PT and by treatment, cohort and overall if considered appropriate.

#### 9.1.2 Local tolerability

An overview of all local tolerability reactions including maximum intensity grade per local tolerability reaction will be presented by part, cohort, treatment, and overall. Intensity grade for each local tolerability reaction will also be presented by cohort, treatment, and overall using a frequency table. Changes from baseline in intensity grade at each time point will be summarised in a shift table.

#### 9.1.3 Vital signs

Vital signs will be summarised by treatment and cohort, and by assessment time point. Data will be presented with absolute and percent change from baseline. Vital signs data (blood pressure and pulse) for eligibility (screening) in Part B will only be listed.

#### 9.1.4 Electrocardiogram

All ECGs will be categorised as "normal", "abnormal, not clinically significant", or "abnormal, clinically significant" (as judged by the Investigator) and summarised by treatment and cohort, and by assessment time point using frequency tables. Changes over time will be presented using a shift table if considered appropriate. All measured ECG values will be summarised by treatment, cohort and overall, and assessment timepoint with absolute and percent change from baseline. ECG data for eligibility (screening) in Part B will only be listed.

#### 9.1.5 Safety laboratory

Safety laboratory data will be summarised by treatment and cohort, and by assessment time point with absolute and percent change from baseline.

All safety laboratory measurements will be categorised as "normal", "abnormal, not clinically significant", or "abnormal, clinically significant" (as judged by the Investigator) and

summarised by treatment and cohort, and by assessment time point using frequency tables. Safety laboratory data for eligibility (screening) in Part B will only be listed.

#### 9.1.6 Physical examinations

Normal and clinically significant and non-clinically significant abnormal findings will be specified and summarised by treatment and cohort, and by assessment time point. Changes over time will be presented using shift tables, if appropriate. Physical examination data for eligibility (screening) in Part B will only be listed.

#### 9.1.7 Cream absorption (Part B)

Cream absorption measured on a 4-point scale will be presented using a frequency table by cohort. The time until adequate abruption, measured at 30 min, 1h, and 2 h, will be presented by cohort in the same frequency table. Adequate abruption will be interpreted as equivalent to a cream absorption score of at least "3 = Mostly absorbed" on the 4-point cream absorption scale.

#### 9.2 Analysis of secondary endpoints

#### 9.2.1 Pharmacokinetic analysis (Part A)

The following non-compartmental plasma PK parameters will be determined/calculated (if data permits) during the trial conduct:

- $T_{max}$  Time to reach  $C_{max}$
- C<sub>max</sub> The maximum observed plasma concentration
- AUC<sub>0-last</sub> Area under the plasma concentration versus time curve (AUC) from timepoint 0 to t, where t represents the timepoint of the last detectable plasma concentration
- AUC<sub>0-inf</sub> AUC from timepoint 0 extrapolated to infinity
- $T_{1/2}$  Terminal plasma elimination half-life

#### Parameters that are only presented in listings

- Lambda<sub>z</sub> Eliminate rate constant associated with the terminal phase
- Lambda<sub>z</sub> lower Lower limit on time for values to be included in the calculation of Lambda<sub>z</sub>
- Lambda<sub>z</sub> upper Upper limit on time for values to be included in the calculation of Lambda<sub>z</sub>
- No points lambda<sub>z</sub> Number of points used in computing lambda<sub>z</sub>
- Span The ratio between the interval used for determination of lambda<sub>z</sub> and the terminal  $T_{1/2}$
- Rsq adj Goodness of fit statistic for the terminal phase, adjusted for the number of points used in the estimation of lambda<sub>Z</sub>.
- AUC<sub>extr</sub>% Percentage of AUC<sub>0-inf</sub> due to extrapolation from T<sub>last</sub> to infinity
- T<sub>last</sub> Last observed concentration

#### Following units will be used:

• Time: h

• Concentration: nmol/L

• AUCs: h\* nmol/L

• Lambda<sub>z</sub>: /h

Non-compartmental analysis will be based on the actual sampling times recorded during the trial.. For the purpose of calculating PK parameters, concentrations below lower limit of quantification (LLOQ) occurring before  $C_{max}$  will be treated as zero. Concentrations below LLOQ occurring after  $C_{max}$  will be omitted from the analysis.

T<sub>max</sub>, T<sub>last</sub> and C<sub>max</sub> will be based on the observed plasma concentration data.

All AUC will be assessed by integration of the plasma concentration vs time curve using linear interpolation for increasing plasma levels and logarithmic interpolation for decreasing plasma levels (Linear Up-Log Down method).

AUC<sub>0-last</sub> will be calculated from time 0 to the time t of the last detectable plasma concentration.

For AUC<sub>0-inf</sub> the area will be calculated to the last timepoint showing a measurable plasma concentration and then extrapolated to infinity using the concentration in the last quantifiable sample and lambda<sub>z</sub>.

$$AUC_{0-inf} = AUC_{0-last} + \frac{C_{last}}{lambda_z}$$

Formulas for calculation of AUC

• Linear trapezoidal rule:

$$AUC|_{t1}^{t2} = \delta t \times \frac{C_1 + C_2}{2}$$

• Logarithmic trapezoidal rule:

$$AUC|_{t1}^{t2} = \delta t \times \frac{C_2 - C_1}{C_2}$$
$$ln(C_1)$$

where t = time, c = concentration,  $\delta t = t_2 - t_1$ .

Formulas for interpolation (to find C\* at time t\* for  $t1 < t^* < t2$ )

• Linear interpolation rule:

$$C^* = C_1 + \left| \frac{t^* - t_1}{t_2 - t_1} \right| (C_2 - C_1)$$

• Logarithmic interpolation rule:

$$C^* = exp \left( ln(C_1) + \left| \frac{t^* - t_1}{t_2 - t_1} \right| * \left( ln(C_2) - ln(C_1) \right) \right)$$

where t = time, c = concentration

Lambda<sub>z</sub>, the first order rate constant associated with the terminal portion of the curve will be determined by lin-logarithmic regression of the terminal elimination phase of individual plasma concentration vs time curves. Determination of lambda<sub>z</sub> requires identification of a sufficiently linear terminal phase (as determined by visual inspection of the lin-log plasma concentration vs time plot with the regression line) consisting of at least 3 terminal concentration values (not including  $C_{max}$ ). If this is not achieved, lambda<sub>z</sub> and its dependent PK parameters will not be reported for that profile.

In the following cases, lambda<sub>z</sub> dependent PK parameters will be flagged in listings as potentially unreliable:

- Lambda<sub>z</sub> estimation is based on a period of less than 1.5 times the resulting  $T_{1/2}$ .
- The Rsq adjusted value of the regression line is < 0.85.
- The estimated % extrapolated AUC is  $\geq 20\%$  ((AUC<sub>0-inf</sub>-AUC<sub>0-last</sub>/AUC<sub>0-inf</sub>)\*100).

 $T_{1/2}$  will be calculated accordingly:

$$T_{1/2} = \frac{\ln(2)}{lambda_z}$$

Span will be calculated accordingly:

$$Span = \frac{lambda_z \; upper - \; lambda_z \; lower}{T_{1/2}}$$

If there is a confirmed dosing error during the trial, the pharmacokinetic data for that period will only be included in the listings but excluded from descriptive and statistical analyses. In case of missed blood samples, potential impact on PK parameters will be assessed for each individual case. PK parameters with a high degree of uncertainty due to missing samples (e.g., multiple samples missing around  $C_{max}$ ) will be flagged as unreliable in the report and may in rare cases be excluded from summary tables, descriptive statistics, and statistical analysis.

### 9.3 Description of trial population

## 9.3.1 Disposition

A participant disposition will be presented by part, showing the number of screened participants; the number of withdrawn participants prior to dose, including the reason for withdrawal; the number of included participants in each cohort; the number of withdrawn participants, including the reason for withdrawal; the number of completed participants; the number of participants included in the analysis sets, and the number of participants at each visit.

## 9.3.2 Demographics and baseline characteristics

Descriptive statistics for demographics, weight and height will be presented for all participants, by part.

#### 9.3.3 Medical/surgical history and prior/concomitant medication

Medical/surgical history will be presented by part, system organ class (SOC) and preferred term (PT). Prior/concomitant medications will be presented by ATC level 4 and WHODrug Preferred name.

## 9.3.4 Investigational medicinal product use

Individual IMP use will be listed.

24(66)

#### 10 DATA DISPLAY PLAN

Tables and figures will only be generated if sufficient data, with sufficient variability exist to justify specific output being produced. Unscheduled/extra visits will generally not be presented in tables and summary figures but will be included in listings.

#### **10.1** Table of contents DDP

| 10.2 | Trial | tables | 27 |
|------|----------|-----------------------------------|----|
| 10. | 2.1 | Demographic data | 27 |
| 10. | 2.2 | Primary endpoints | 37 |
| 1 | 10.2.2.1 | Adverse events | 37 |
| 1 | 10.2.2.2 | Local tolerability | 42 |
| 1 | 10.2.2.3 | Vital signs (Part A) | 49 |
| 1 | 10.2.2.4 | 12-lead ECG (Part A) | 50 |
| 1 | 10.2.2.5 | Safety laboratory (Part A) | 53 |
| 1 | 10.2.2.6 | Physical examinations (Part A) | 55 |
| 1 | 10.2.2.7 | Cream absorption (Part B) | 57 |
| 10. | 2.3 | Secondary endpoints (Part A) | 58 |
| 1 | 10.2.3.1 | Pharmacokinetic analysis (Part A) | 58 |
| 10.3 | Trial | figures | 60 |
| 10. | 3.1 | Secondary endpoints (Part A) | 60 |
| | 10.3.1.1 | Pharmacokinetic analysis (Part A) | 60 |
| 10.4 | Trial | listings | 64 |

| List | of | tabl | es |
|------|----|------|----|
|------|----|------|----|

| Table DM 1 | Baseline characteristics and demographics - Part A (Full analysis set) | 27 |
|---|---|---|
| Table DM 2 | Baseline characteristics and demographics - Part B (Full analysis set) | 28 |
| Table DS 1 | Participant disposition – Part A (All participants) | 30 |
| Table DS 2 | Participant disposition – Part B (All participants) | 31 |
| Table MH 1<br>(Full analysis se | Medical history events by system organ class and preferred term – Part A et) | 32 |
| Table MH 2<br>(Full analysis se | Medical history events by system organ class and preferred term – Part B et) | 32 |
| Table CM 1<br>analysis set) | Prior medications by ATC level 4 and preferred name – Part A (Full 33 | |
| Table CM 2 set) | Prior medications by ATC level 4 and preferred name – Part B (Full analy 34 | /sis |
| Table CM 3 analysis set) | Concomitant medications by ATC level 4 and preferred name – Part A (F 35 | ull |
| Table CM 4<br>analysis set) | Concomitant medications by ATC level 4 and preferred name – Part B (Fig. 36) | ull |
| Table AE 1 | Overview of adverse events – Part A (Full analysis set) | 37 |
| Table AE 2 | Overview of adverse events – Part B (Full analysis set) | 38 |
| Table AE 3 analysis set) | Adverse events by system organ class and preferred term – Part A (Full 39 | |
| Table AE 4<br>analysis set) | Adverse events by system organ class and preferred term – Part B (Full $40$ | |
| Table AE 5<br>(Full analysis se | Serious adverse events by system organ class and preferred term – Part A et) | 41 |
| Table AE 6<br>(Full analysis se | Serious adverse events by system organ class and preferred term – Part B et) | 41 |
| Table AE 7 Tre<br>A (Full analysis | atment related adverse events by system organ class and preferred term – P s set) | art<br>41 |
| Table AE 8 Tre<br>B (Full analysis | atment related adverse events by system organ class and preferred term – P set) | art<br>41 |
| Table LT 1 | Overview of local tolerability – Part A (Full analysis set) | 42 |
| Table LT 2 | Overview of local tolerability – Part B (Full analysis set) | 44 |
| Table LT 3 | Local tolerability intensity grades – Part A (Full analysis set) | 46 |
| Table LT 4 | Local tolerability intensity grades – Part B (Full analysis set) | 47 |
| Table LT 5 | Local tolerability intensity grades shift table – Part A (Full analysis set) | 47 |
| Table LT 6 | Local tolerability intensity grades shift table – Part B (Full analysis set) | 48 |


| Table LB 1 set) | Safety laboratory measurements: Clinical chemistry – Part A (Full analyst 53 | is |
|---|---|---|
| Table LB 2 set) | Safety laboratory interpretations: Clinical chemistry – Part A (Full analys 54 | is |
| Table LB 3 | Safety laboratory measurements: Haematology - Part A (Full analysis set | )55 |
| Table LB 4 | Safety laboratory interpretations: Haematology – Part A (Full analysis set 55 | t) |
| Table LB 5 | Safety laboratory measurements: Coagulation - Part A (Full analysis set) | 55 |
| Table LB 6 | Safety laboratory interpretations: Coagulation - Part A (Full analysis set) | 55 |
| Table VS 1 | Vital signs measurements – Part A (Full analysis set) | 49 |
| Table EG 1 | ECG measurements – Part A (Full analysis set) | 50 |
| Table EG 2 | ECG interpretations – Part A (Full analysis set) | 51 |
| Table EG 3 | ECG interpretations shift table – Part A (Full analysis set) | 52 |
| Table PE 1 | Physical examinations – Part A (Full analysis set) | 55 |
| Table PE 2 | Physical examinations shift table – Part A (Full analysis set) | 56 |
| Table QS 1 | Cream absorption – Part B (Full analysis set) | 57 |
| Table PC 1 | Plasma concentrations – Part A (Pharmacokinetic analysis set) | 58 |
| Table PP 1 | PK parameters – Part A (Pharmacokinetic analysis set) | 58 |
| List of figures | | |
| Figure PC 1 (Pharmacokine | Geometric mean plasma concentrations over time (lin-log) – Part A tic analysis set) | 60 |
| Figure PC 2 (Pharmacokine | Geometric mean plasma concentrations over time (lin-lin) – Part A tic analysis set) | 61 |
| Figure PC 3 set) | Individual plasma concentrations over time (lin-log) – Part A (Full analys 61 | is |
| Figure PC 4 set) | Individual plasma concentrations over time (lin-lin) – Part A (Full analysi 63 | is |


## 10.2 Trial tables

## 10.2.1 Demographic data

Table DM 1 Baseline characteristics and demographics – Part A (Full analysis set)

| Assessment (unit) | | | | | | | |
|---|---|---|---|---|---|---|---|
| Age (years) | n | x | х | х | х | х | Х |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Min, Max) | xx.x (xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) |
| Height (cm) | n | x | х | х | х | х | Х |
| | Mean (SD) | xxx.x (xx.x) | xxx.x (xx.x) | xxx.x (xx.x) | xxx.x (xx.x) | xxx.x (xx.x) | xxx.x (xx.x) |
| | Median (Min, Max) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) |
| Weight (kg) | n | x | х | х | х | х | х |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) |
| Body Mass Index (kg/m2) | n | x | x | x | x | x | х |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx(xx.x,xx.x) |
| BSA (m2) | n | x | х | х | х | х | х |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) | xx.xx(xx.x,xx.x) | xx.xx (xx.x, xx.x) | xx.xx(xx.x,xx.x) | xx.xx (xx.x, xx.x) | xx.xx(xx.x,xx.x) |
| Sex | Female | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Male | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Ethnicity | Hispanic or latino | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not hispanic or latino | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not reported | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | | • | | | | | |


| Assessment (unit) | | | | | | | |
|---|---|---|---|---|---|---|---|
| | Unknown | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Race | American Indian or Alaska Native | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Asian | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Black or African American | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Native Hawaiian or Other Pacific Islander | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | White | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in treatment group. Percentages are based on the number of observations. n: Number of observations. SD: Standard deviation. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table DM 2 Baseline characteristics and demographics -

| Age (years) | n | x | X | X | X |
|---|---|---|---|---|---|
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| - | Median (Min, Max) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) |
| Height (cm) | n | x | X | X | X |
| | Mean (SD) | xxx.x (xx.x) | xxx.x (xx.x) | xxx.x (xx.x) | xxx.x (xx.x) |
| | Median (Min, Max) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) |
| Weight (kg) | n | X | х | X | X |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) |
| Body Mass Index (kg/m2) | n | x | х | X | Х |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) |


#### **Ankh Life Sciences Limited**

Statistical Analysis Plan A24-0001 Final v4.0

| Assessment (unit) | | | | | |
|---|---|---|---|---|---|
| BSA (m2) | n | х | X | X | Х |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) | xx.xx (xx.x, xx.x) | xx.xx(xx.x,xx.x) | xx.xx(xx.x,xx.x) |
| Sex | Female | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Male | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Ethnicity | Hispanic or latino | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not hispanic or latino | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not reported | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Unknown | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Race | American Indian or Alaska Native | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Asian | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Black or African American | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Native Hawaiian or Other Pacific Islander | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | White | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in treatment group. Percentages are based on the number of observations. n: Number of observations. SD: Standard deviation. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


Table DS 1 Participant disposition – Part A (All participants)

| | Total<br>(N=XXX) |
|------------------------------------------|------------------|
| Screened participants | xxx |
| Withdrawn prior to dose | xxx |
| Reason for withdrawal prior to dose | |
| Reason 1 | xxx |
| Reason 2 | xxx |
| <del></del> | xxx |
| Participants included in trial | xxx |
| Allocated to arm | |
| | xxx |
| | xxx |
| | xxx |
| | xxx |
| | xxx |
| Withdrawn participants | |
| Reason 1 | xxx |
| Reason 2 | XXX |
| <del></del> | XXX |
| Completed participants | XXX |
| Included in Full analysis set | XXX |
| Included in Pharmacokinetic analysis set | xxx |
| Participants at each visit | |
| Visit 1 - Screening | xxx |
| Visit 2 - Inpatient stay | xxx |
| Visit 3 - Follow-up | xxx |

Data based on All participants. BSA: Body surface area. ¹The data for participants receiving placebo is presented pooled across groups. SAS program: [PROGRAM NAME].sas. Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


**Table DS 2** Participant disposition – Part B (All participants)

| | Total<br>(N=XXX) |
|-------------------------------------|------------------|
| Screened participants | xxx |
| Withdrawn prior to dose | xxx |
| Reason for withdrawal prior to dose | |
| Reason 1 | XXX |
| Reason 2 | XXX |
| <del></del> | XXX |
| Participants included in trial | XXX |
| Allocated to arm | |
| | XXX |
| | XXX |
| | XXX |
| Withdrawn participants | |
| Reason 1 | XXX |
| Reason 2 | XXX |
| <del></del> | XXX |
| Completed participants | XXX |
| Included in Full analysis set | XXX |
| Participants at each visit | |
| Visit 1 - Screening | XXX |
| Visit 2 – Treatment visit | XXX |
| Visit 3 - Follow-up | xxx |

Data based on All participants. BSA: Body surface area. SAS program: [PROGRAM NAME].sas. Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


Table MH 1 Medical history events by system organ class and preferred term – Part A (Full analysis set)

| System organ class | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred term | | | | | | | | | | | | m |
| Total | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 1 PT 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 1 PT 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
| [SOC 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [SOC 2 PT 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 2 PT 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2 PT] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [SOC] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [SOC PT 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [SOC PT 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX |
| [SOC PT] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following events are coded with multiple terms and are represented as separate events in tables and listings: '[MH TERM 1], [MH TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table MH 2 Medical history events by system organ class and preferred term – Part B (Full analysis set)

| System organ class Preferred term | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Total | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | _ |


| | | | | | | | | <u> </u> |
|---|---|---|---|---|---|---|---|---|
| System organ class<br>Preferred term | | | | | | | | m |
| [SOC 1] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [SOC 1 PT 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT 2] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [SOC 2 PT 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2 PT 2] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2 PT] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [SOC PT 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC PT 2] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC PT] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following events are coded with multiple terms and are represented as separate events in tables and listings: '[MH TERM 1], [MH TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table CM 1 Prior medications by ATC level 4 and preferred name – Part A (Full analysis set)

| | | | | | | | | | | | Total<br>(N=XX) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ATC Name Level 4<br>Preferred Name | | | | | | | | | | m | n (%) | m |
| Total | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
| [L4 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 1 PN 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |


| | | | | | | | | | | | _ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | Total<br>(N=XX) | |
| ATC Name Level 4 Preferred Name | n (%) | m | n (%) | m | n (%) | m | n (%) | m | n (%) | m | n (%) | m |
| [L4 1 PN 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 1 PN] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 2 PN 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 2 PN 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 2 PN] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 PN 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 PN 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 PN] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following records are coded with multiple terms and are represented as separate events in tables and listings: '[CM TERM 1], [CM TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table CM 2 Prior medications by ATC level 4 and preferred name – Part B (Full analysis set)

| ATC Name Level 4 Preferred Name | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|
| Total | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 1 PN 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 1 PN 2] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 1 PN] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |


| ATC Name Level 4<br>Preferred Name | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|
| [L4 2] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 2 PN 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 2 PN 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 2 PN] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 PN 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 PN 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 PN] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following records are coded with multiple terms and are represented as separate events in tables and listings: '[CM TERM 1], [CM TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas
Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table CM 3 Concomitant medications by ATC level 4 and preferred name – Part A (Full analysis set)

| | | | | | | | | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ATC Name Level 4<br>Preferred Name | | | | | | | | | | m | (N=XX)<br>n (%) | m |
| Total | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [L4 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 1 PN 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [L4 1 PN 2] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [L4 1 PN] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [L4 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [L4 2 PN 1] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |

| | | | | | | | | | | | _ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | Total<br>(N=XX) | |
| ATC Name Level 4 Preferred Name | | | | | | | | | | m | n (%) | m |
| [L4 2 PN 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [L4 2 PN] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 PN 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [L4 PN 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [L4 PN] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following records are coded with multiple terms and are represented as separate events in tables and listings: '[CM TERM 1], [CM TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table CM 4 Concomitant medications by ATC level 4 and preferred name – Part B (Full analysis set)

| ATC Name Level 4 Preferred Name | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|
| Total | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 1 PN 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 1 PN 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 1 PN] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 2 PN 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 2 PN 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [L4 2 PN] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |


| | | | | | | _ | | |
|---|---|---|---|---|---|---|---|---|
| ATC Name Level 4 | | | | | | | | |
| Preferred Name | | | | | | | | m |
| [L4] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 PN 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 PN 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [L4 PN] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following records are coded with multiple terms and are represented as separate events in tables and listings: '[CM TERM 1], [CM TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

# 10.2.2 Primary endpoints

#### 10.2.2.1 Adverse events

Table AE 1 Overview of adverse events – Part A (Full analysis set)

| Any AE | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Any SAE | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Any AE leading to withdrawal from trial | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Any AE leading to death | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Causality | | | | | | | | | | | | |
| Not related | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Unlikely related | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Possibly related | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |


| | | | | | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Probably related | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Definitely related | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| Severity | | | | | | | | | | | | |
| Mild | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Moderate | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Severe | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Life-Threatening | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Death | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following AEs are coded with multiple MedDRA terms and are represented as separate AEs in tables and listings: '[AE TERM 1]', '[AE TERM 2]', '[AE TERM 3]. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

**Table AE 2** Overview of adverse events – Part




| Probably related | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
|---|---|---|---|---|---|---|---|---|
| Definitely related | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Severity | | | | | | | | |
| Mild | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Moderate | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Severe | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Life-Threatening | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Death | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following AEs are coded with multiple MedDRA terms and are represented as separate AEs in tables and listings: '[AE TERM 1]', '[AE TERM 2]', '[AE TERM 3]. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table AE 3 Adverse events by system organ class and preferred term – Part A (Full analysis set)

| System organ class<br>Preferred term | n (%) | m | n (%) | m | n (%) | m | n (%) | m | n (%) | m | n (%) | m |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Total | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [SOC 1] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [SOC 1 PT 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| [SOC 1 PT 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 1 PT] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 2 PT 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 2 PT 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |


| | | | _ | | | | | | | | _ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System organ class<br>Preferred term | | | | | | | | | | | | |
| [SOC 2 PT] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [SOC] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [SOC PT 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
| [SOC PT 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
| [SOC PT] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following events are coded with multiple terms and are represented as separate events in tables and listings: '[AE TERM 1], [AE TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table AE 4 Adverse events by system organ class and preferred term – Part B (Full analysis set)

| System organ class Preferred term | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|
| Total | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
| [SOC 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX |
| [SOC 2 PT 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2 PT 2] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2 PT] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |


| System organ class | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred term | | | | | | | | m |
| [SOC PT 1] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC PT 2] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC PT] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. The following events are coded with multiple terms and are represented as separate events in tables and listings: '[AE TERM 1], [AE TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

## Table AE 5 Serious adverse events by system organ class and preferred term – Part A (Full analysis set)

Same layout as Table AE 3

# Table AE 6 Serious adverse events by system organ class and preferred term – Part B (Full analysis set)

Same layout as Table AE 4

### Table AE 7 Treatment related adverse events by system organ class and preferred term – Part A (Full analysis set)

Same layout as Table AE 3. Add footnote: An AE is considered causally related to the use of the IMP when the causality assessment is probably, possibly or definitely related.

### Table AE 8 Treatment related adverse events by system organ class and preferred term – Part B (Full analysis set)

Same layout as Table AE 4. Add footnote: An AE is considered causally related to the use of the IMP when the causality assessment is probably, possibly or definitely related.


# 10.2.2.2 Local tolerability

Table LT 1 Overview of local tolerability – Part A (Full analysis set)

| | | | | , | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | m |
| Any LT reaction graded higher than None | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Any Erythema | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Erythema | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Swelling | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Swelling | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Pruritus | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Pruritus | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Burning | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Burning | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |


| | | | | | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Blistering | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Blistering | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Urticaria | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Urticaria | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Discolouration | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Discolouration | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Dryness | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Dryness | | | | | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |


| | | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|---|
| Moderate | xx (xx%) | xx (xx%) | xx (xx%) | XX | xx (xx%) | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | xx (xx%) | xx (xx%) | XX | xx (xx%) | xx (xx%) | XX | xx (xx%) | |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table LT 2 Overview of local tolerability – Part B (Full analysis set)

| | | | | | | | | m |
|---|---|---|---|---|---|---|---|---|
| Any LT reaction graded higher than None | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Any Erythema | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
| Maximum grade Erythema | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Swelling | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Swelling | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |
| Any Pruritus | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Pruritus | | | | | | | | |


| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
|---|---|---|---|---|---|---|---|---|
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Burning | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Burning | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Blistering | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Blistering | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Any Urticaria | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX |
| Maximum grade Urticaria | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |
| Any Discolouration | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | xx |
| Maximum grade Discolouration | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |


| | | | | | | | _ | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | | m |
| Moderate | xx (xx%) | | xx (xx%) | · | xx (xx%) | xx | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |
| Any Dryness | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |
| Maximum grade Dryness | | | | | | | | |
| None | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |
| Mild | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |
| Moderate | xx (xx%) | | xx (xx%) | | xx (xx%) | xx | xx (xx%) | |
| Severe | xx (xx%) | | xx (xx%) | | xx (xx%) | XX | xx (xx%) | |

Data based on [ANALYSIS SET]. BSA: Body surface area. N: number of participants in the treatment group. Percentages are based on N. n: number of participants. m: number of events. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table LT 3 Local tolerability intensity grades – Part

| [PARAMETER 1] | [Assessment timepoint 1] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
|---|---|---|---|---|---|---|---|---|
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [Assessment timepoint 2] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Data based on [population]. SAS program: [PROGRAM NAME].sas. BSA: Body surface area. N: Number of participants in the treatment group. Percentages are based on the number of observations.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


Table LT 4 Local tolerability intensity grades – Part B (Full analysis set)

| Assessment | Assessment timepoint | | | | | |
|---|---|---|---|---|---|---|
| [PARAMETER 1] | [Assessment timepoint 1] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [Assessment timepoint 2] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table LT 5 Local tolerability intensity grades shift table – Part A (Full analysis set)

| Parameter | Assessment timepoint | Baseline value | Post-baseline value | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | [BASELINE] | [RESPONSE 1] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 1] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX(xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX(xx%) | xx/XX (xx%) | xx/XX(xx%) | xx/XX(xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |


| Parameter | Assessment timepoint | Baseline value | Post-baseline value | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 2] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX(xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table LT 6 Local tolerability intensity grades shift table – Part B (Full analysis set)

| Parameter | Assessment timepoint | Baseline value | | | | | |
|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | [BASELINE] | [RESPONSE 1] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 1] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |


| Parameter | Assessment timepoint | Baseline value | Post-baseline value | | | | |
|---|---|---|---|---|---|---|---|
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 2] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

# 10.2.2.3 Vital signs (Part A)

Table VS 1 Vital signs measurements – Part A (Full analysis set)

| Assessment (unit) | Result category | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | Measured value | [Assessment | n | xx | XX | XX | XX | XX |
| (unit) | | timepoint 1] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |


| Assessment (unit) | Result category | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx (x.x, x.x) |
| | | [Assessment | n | xx | xx | xx | xx | XX |
| | | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Change from | [Assessment | n | xx | xx | xx | XX | XX |
| | baseline | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Relative change from | [Assessment | n | xx | xx | xx | xx | XX |
| | baseline (%) | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |

Data based on [population]. BSA: Body surface area. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. IQR: Inter-quartile range. Q1: Lower quartile. Q3: Upper quartile. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

# 10.2.2.4 12-lead ECG (Part A)

Table EG 1 ECG measurements – Part A (Full analysis set)

| Assessment (unit) | Result category | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | Measured value | [Assessment | n | xx | XX | XX | XX | XX |
| (unit) | | timepoint 1] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |


| Assessment (unit) | Result category | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| | | [Assessment | n | xx | xx | xx | xx | xx |
| | | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Change from baseline | [Assessment | n | xx | XX | XX | XX | XX |
| | baseline | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Relative change from baseline (%) | | n | xx | XX | XX | xx | XX |
| | baseline (%) | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |

Data based on [population]. BSA: Body surface area. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. IQR: Inter-quartile range. Q1: Lower quartile. Q3: Upper quartile. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table EG 2 ECG interpretations – Part A (Full analysis set)

| Assessment | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | [Assessment timepoint 1] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |


| Assessment | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|
| | [Assessment timepoint 2] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table EG 3 ECG interpretations shift table – Part A (Full analysis set)

| Parameter | Assessment timepoint | Baseline value | Post-baseline value | | | | | |
|---|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | [BASELINE] | [RESPONSE 1] | NA | xx/XX (xx%) | xx/XX(xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | NA | xx/XX (xx%) | xx/XX(xx%) | xx/XX ( $xx%$ ) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | NA | xx/XX (xx%) | xx/XX(xx%) | xx/XX(xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 1] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX(xx%) | xx/XX(xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX(xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX(xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX(xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 2] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |


| Parameter | Assessment timepoint | Baseline value | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

# 10.2.2.5 Safety laboratory (Part A)

Table LB 1 Safety laboratory measurements: Clinical chemistry – Part A (Full analysis set)

| Assessment (unit) | Result category | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|---|
| [PARAMETER 1] (unit) | Measured value | [Assessment timepoint 1] | n | | | | | |
| (unit) | | timepoint 1 | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | | [Assessment | n | xx | xx | xx | xx | XX |
| | | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, x.x) |


| Assessment (unit) | Result category | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|---|
| <u> </u> | Change from | [Assessment | n | xx | xx | xx | xx | xx |
| | baseline | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| | Relative change from | | n | xx | xx | xx | xx | xx |
| | baseline (%) | timepoint 2] | n/BLQ/ULQ | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx | xx/xx/xx |
| | | | Mean (SD | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, x.x) |

Data based on [population]. BSA: Body surface area. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. IQR: Inter-quartile range. Q1: Lower quartile. Q3: Upper quartile. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table LB 2 Safety laboratory interpretations: Clinical chemistry – Part A (Full analysis set)

| Assessment | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | [Assessment timepoint 1] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [Assessment timepoint 2] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Data based on [population]. SAS program: [PROGRAM NAME].sas. BSA: Body surface area.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


### Table LB 3 Safety laboratory measurements: Haematology – Part A (Full analysis set)

Same layout as Table LB 1

### Table LB 4 Safety laboratory interpretations: Haematology – Part A (Full analysis set)

Same layout as Table LB 2

### Table LB 5 Safety laboratory measurements: Coagulation – Part A (Full analysis set)

Same layout as Table LB 1

#### Table LB 6 Safety laboratory interpretations: Coagulation – Part A (Full analysis set)

Same layout as Table LB 2

### 10.2.2.6 Physical examinations (Part A)

Table PE 1 Physical examinations – Part A (Full analysis set)

| Assessment | Assessment timepoint | | | | | | |
|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | [Assessment timepoint 1] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [Assessment timepoint 2] | [RESULT 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESULT 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Data based on [population]. SAS program: [PROGRAM NAME].sas. BSA: Body surface area. N: Number of participants in the treatment group. Percentages are based on the number of observations.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


Table PE 2 Physical examinations shift table – Part A (Full analysis set)

| Parameter | Assessment timepoint | Baseline value | Post-baseline value | | | | | |
|---|---|---|---|---|---|---|---|---|
| [PARAMETER 1] | [BASELINE] | [RESPONSE 1] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | NA | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 1] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [POST BASELINE 2] | [RESPONSE 1] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 2] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | [RESPONSE 3] | [RESPONSE 1] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 2] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | | [RESPONSE 3] | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


# 10.2.2.7 Cream absorption (Part B)

Table QS 1 Cream absorption – Part B (Full analysis set)

| Assessment (unit) | Assessment timepoint | | | | |
|---|---|---|---|---|---|
| Cream absorption | [Assessment timepoint 1] | 1= Not absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 2= Somewhat absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 3= Mostly absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 4= Completely absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [Assessment timepoint 2] | 1= Not absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 2= Somewhat absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 3= Mostly absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 4= Completely absorbed | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| Time until adequate abruption (unit) | [Assessment timepoint 1] | 30 min | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 1 h | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 2 h | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | [Assessment timepoint 2] | 30 min | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 1 h | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |
| | | 2 h | xx/XX (xx%) | xx/XX (xx%) | xx/XX (xx%) |

Data based on [population]. SAS program: [PROGRAM NAME].sas. Adequate abruption is interpreted as equivalent to a cream absorption score of at least "3 = Mostly absorbed" on the 4-point cream absorption scale. BSA: Body surface area N: Number of participants in the treatment group. n: Number of observations.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


# 10.2.3 Secondary endpoints (Part A)

# 10.2.3.1 Pharmacokinetic analysis (Part A)

Table PC 1 Plasma concentrations – Part A (Pharmacokinetic analysis set)

| Assessment (unit) | Assessment timepoint | | | | | |
|---|---|---|---|---|---|---|
| [PARAMETER 1] (unit) | [Assessment timepoint 1] | n/BLQ | xx/xx | xx/xx | xx/xx | xx/xx |
| | | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| | [Assessment timepoint 2] | n/BLQ | xx/xx | xx/xx | xx/xx | xx/xx |
| | | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |

Data based on [population]. BSA: Body surface area. LLOQ is xx (unit). See listing 16.2.5-1 for a per participant LLOQ summary. n: Number of observations. BLQ: Below lower limit of quantification. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3 or more than half of the observations are BLQ. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Table PP 1 PK parameters – Part A (Pharmacokinetic analysis set)

| Assessment (unit) | | | | | |
|---|---|---|---|---|---|
| Tmax (unit) | n | xx | XX | XX | XX |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |


| Assessment (unit) | | | | | |
|---|---|---|---|---|---|
| max (unit) | n | XX | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| AUC0-last (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx(x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| UC0-inf (unit) | n | xx | XX | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| T1/2 (unit) | n | xx | XX | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |

Data based on [population].: Body surface area. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3 or more than half of the observations are BLQ. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas.

Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


## 10.3 Trial figures

### 10.3.1 Secondary endpoints (Part A)

# 10.3.1.1 Pharmacokinetic analysis (Part A)

Figure PC 1 Geometric mean plasma concentrations over time (lin-log) – Part A (Pharmacokinetic analysis set)



Example figure. Note that the numbers do not reflect real data. This template figure will be adjusted as needed depending on the collected data.

Data based on [population]. BSA: Body surface area. Individual values under LLOQ are excluded from the figure. LLOQ is xx (unit). See listing 16.2.5-1 for a per participant LLOQ summary. SAS program: [PROGRAM NAME].sas. Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.




Figure PC 2 Geometric mean plasma concentrations over time (lin-lin) – Part A (Pharmacokinetic analysis set)

Example figure. Note that the numbers do not reflect real data. This template figure will be adjusted as needed depending on the collected data.

Data based on [population]. BSA: Body surface area. Individual values under LLOQ are excluded from the figure. LLOQ is xx (unit). See listing 16.2.5-1 for a per participant LLOQ summary. SAS program: [PROGRAM NAME].sas. Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.

Figure PC 3 Individual plasma concentrations over time (lin-log) – Part A (Full analysis set)

Individual values under LLOQ will be excluded from the figure.




Example figure. Note that the numbers do not reflect real data. This template figure will be adjusted as needed depending on the collected data.

Data based on [population]. BSA: Body surface area. Individual values under LLOQ are excluded from the figure. LLOQ is xx (unit). See listing 16.2.5-1 for a per participant LLOQ summary. SAS program: [PROGRAM NAME].sas. Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


Figure PC 4 Individual plasma concentrations over time (lin-lin) – Part A (Full analysis set)

Individual values under LLOQ will be excluded from the figure.



Example figure. Note that the numbers do not reflect real data. This template figure will be adjusted as needed depending on the collected data.

Data based on [population]. BSA: Body surface area. Individual values under LLOQ are excluded from the figure. LLOQ is xx (unit). See listing 16.2.5-1 for a per participant LLOQ summary. lin: Linear. SAS program: [PROGRAM NAME].sas. Dataset version: ADXX YYYY-MM-DDTHH:MM:SS. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. EDC data extracted: YYYY-MM-DDTHH:MM:SS.


#### **10.4** Trial listings

### 16.2.1 Discontinued participants

- Listing 16.2.1-1 Discontinued participants Part A
- Listing 16.2.1-2 Discontinued participants Part B
- Listing 16.2.1-3 Non-eligible participants Part A
- Listing 16.2.1-4 Non-eligible participants Part B
- Listing 16.2.1-5 Disposition Part A (All participants)
- Listing 16.2.1-6 Disposition Part B (All participants)
- Listing 16.2.1-7 Participant visits Part A (All participants)
- Listing 16.2.1-8 Participant visits Part B (All participants)
- Listing 16.2.1-9 Participant elements Part A (All participants)
- Listing 16.2.1-10 Participant elements Part B (All participants)

#### 16.2.2 Protocol deviations

- Listing 16.2.2-1 Protocol deviations Part A (All participants)
- Listing 16.2.2- 2 Protocol deviations Part B (All participants)

### 16.2.3 Participants excluded from the analysis

- Listing 16.2.3-1 Population definitions Part A (All participants)
- Listing 16.2.3-2 Population definitions Part B (All participants)

#### 16.2.4 Demographic data


- Listing 16.2.4-1 Demography Part A (All participants)
- Listing 16.2.4- 2 Demography Part B (All participants)
- Listing 16.2.4-3 Medical History Part A (All participants)
- Listing 16.2.4-4 Medical History Part B (All participants)
- Listing 16.2.4-5 Prior and concomitant medications Part A (All participants)
- Listing 16.2.4- 6 Prior and concomitant medications Part B (All participants)

#### 16.2.5 Compliance and/or Drug Concentration Data

- Listing 16.2.5-1 Plasma concentration data Part A (All participants)
- Listing 16.2.5-2 Pharmacokinetic parameters Part A (All participants)
- Listing 16.2.5-3 IMP administration Part A (All participants)
- Listing 16.2.5-4 IMP administration Part B (All participants)
- Listing 16.2.5-5 Cream absorption evaluation Part B (All participants)

#### 16.2.6 Individual Efficacy Response Data

NA

### 16.2.7 Adverse event listings (each participant)

- Listing 16.2.7-1 Adverse events Part A (All participants)
- Listing 16.2.7-2 Adverse events Part B (All participants)
- Listing 16.2.7-3 Serious adverse events Part A (All participants)
- Listing 16.2.7-4 Serious adverse events Part B (All participants)

### 16.2.8 Listings of individual laboratory measurements by participant

- Listing 16.2.8-1 Safety laboratory measurements: Clinical chemistry Part A (All participants)
- Listing 16.2.8-2 Safety laboratory measurements: Clinical chemistry Part B (All participants)


- Listing 16.2.8-3 Safety laboratory measurements: Haematology Part A (All participants)
- Listing 16.2.8- 4 Safety laboratory measurements: Haematology Part B (All participants)
- Listing 16.2.8-5 Safety laboratory measurements: Coagulation Part A (All participants)
- Listing 16.2.8- 6 Safety laboratory measurements: Coagulation Part B (All participants)
- Listing 16.2.8-7 Other laboratory measurements Part A (All participants)
  Urine drug screen, alcohol test, pregnancy test
- Listing 16.2.8- 8 Other laboratory measurements Part B (All participants)
  Urine drug screen, alcohol test, pregnancy test
- Listing 16.2.8-9 Virology Part A (All participants)
- Listing 16.2.8- 10 Virology Part B (All participants)

### 16.2.9 Listings of vital signs, ECG, physical examination data by participant

- Listing 16.2.9-1 Vital signs Part A (All participants)
- Listing 16.2.9- 2 Vital signs Part B (All participants)
- Listing 16.2.9-3 ECG Part A (All participants)
- Listing 16.2.9-4 ECG Part B (All participants)
- Listing 16.2.9-5 Physical examinations Part A (All participants)
- Listing 16.2.9- 6 Physical examinations Part B (All participants)
